CLINICAL TRIAL: NCT00686972
Title: The Effect of Surgically Induced Weight Loss on Endocrine Function, Cardiovascular Function and Body Composition
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left JHU
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NA_00004876
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Bariatric Surgery
Keywords: Bariatric Surgery; Glucose Regulation; Cardiac Function; Body Composition
MeSH Terms: interventions — Glucagon-Like Peptide 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GLP-1 (Experimental): 5 ng/kg/min, IV for 1 hour during each clamp study (7) over 2 year period.
  Interventions: Drug: GLP-1

INTERVENTIONS:
Drug: GLP-1 — 5 ng/kg/min, IV for 1 hour during each clamp study (7) over 2 year period.
  Other Names: Glucagon-like Peptide-1

SUMMARY:
This study is being conducted to evaluate changes in sugar, metabolism, heart function and changes in body composition as patients lose weight following bariatric surgery. The investigators will compare improvements of the above changes as a function of the four different types of bariatric surgery. The investigators believe the most beneficial and safest procedure will be the Roux-en-Y.

DETAILED DESCRIPTION:
The study will also examine the response of the pancreas (the insulin-producing organ) to a sugar load, as well as to a hormone called Glucagon Like Peptide 1 (GLP-1), which is released from your gut to maximally stimulate your pancreas. The release of this hormone increases when you eat food and it causes the pancreas to release more insulin than does sugar alone. Volunteers will have 22 visits over a two year period. Only people having Roux-en-Y gastric bypass surgery, gastric sleeve surgery, duodenal switch gastric surgery or lap-band/gastric banding surgery may join. Seventy volunteers will be recruited to take part in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers 21-65 years.
* BMI > 40.
* Preoperative hematocrit level of at least 34% for women and 38% for men.
* Postoperative hematocrit level of at least 34% for women and 36% for men.

Exclusion Criteria:

* Volunteers whose hematocrit level does not meet the above criteria.
* Pregnant and or lactating females.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dariush Elahi, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Glucagon Like Peptide 1 -GLP-1: 5 ng/kg/min, IV for 1 hour during each clamp study (7) over 2 year period.
  GLP-1: 5 ng/kg/min, IV for 1 hour during each clamp study (7) over 2 year period.
Period: Overall Study
Arm/Group | Glucagon Like Peptide 1 -GLP-1
Started | 51
Completed | 0
Not Completed | 51
Not completed — P.I, Left institution. Study terminated | 51

BASELINE CHARACTERISTICS:
Arm/Group | GLP-1
Number analyzed (Participants) | 51
Age, Customized [Number; unit: participants]
  >=21 and <=65 | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Insulin Secretion
Time Frame: 2 years
Population: The PI left the institution and this study was terminated due to noncompliance with our Institutional Review Board. Outcome measure data, if collected, is unknown since no data are available.
Arm/Group | GLP-1
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The PI left the institution and this study was terminated due to noncompliance with our Institutional Review Board. Adverse Event data, if collected, is unknown since no data are available.
Arm/Group | GLP-1
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes